CLINICAL TRIAL: NCT07153107
Title: R01_PilotStudy2_Jaw Muscle Metabolic and Brain-Derived Phenotypes of Chronic TMD Pain
Brief Title: R01_Pilot Jaw Muscle Phenotypes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00025509
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic TMD Pain; Temporomandibular Disorder
Keywords: Jaw Pain; Local Heat Therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-care with local heat therapy (Active Comparator)
  Interventions: Other: Local Heat Therapy
- Self-care without local heat therapy (No Intervention)

INTERVENTIONS:
Other: Local Heat Therapy — This will use a simple device provided to participants named "jaw bra", which is a head wrap with straps that goes around the chin and head that holds heated gel packs over the cheeks area
  Arms: Self-care with local heat therapy

SUMMARY:
The proposed study will assess the effect of local heat therapy on jaw pain and jaw fatigue secondary to a teeth clenching task in chronic TMD pain cases. Researchers expect that most participants will respond to heat therapy and consequently experience reduced jaw pain and fatigue during teeth clenching. The study will assess the clinical characteristics of those participants who respond and do not respond to local heat therapy, in order to determine the common clinical characteristics for those in each response category.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of study participation.
* Be 18 years or older.
* Have a minimum set of teeth present, be it natural, implant-supported or fixed prosthodontics: all anterior teeth (incisors, canines), at least one premolar, at least one molar (first or second molar; third molars not considered).
* TMD-Pain screener score equal to or greater than 3
* Myalgia (masticatory muscle pain) based on clinical exam following the DC/TMD protocol
* Concurrent arthralgia (TMJ pain) and/or headache attributed to TMD allowed
* Myofascial pain must meet the following criteria:

  1. Onset >3 months, occurring >15 days/month on average in the last three months from the screening session
  2. Minimum of 10 jaw pain episodes since onset, each episode lasting at least 30 minutes and no less than 2 hours within the day, OR unremitting

Exclusion Criteria:

* Traumatic facial injury or surgery on the face/jaw, arms or hands;
* Presence of pain related to dental and periodontal pathology;
* Currently undergoing active orthodontic treatment;
* Pregnant;
* Has any of the following medical conditions by self-report:

  1. Renal failure or dialysis,
  2. Heart disease (examples: uncontrolled arrythmia or hypertension, cardiomyopathy) or heart failure, Non-allergic bronchospasm (chronic obstructive pulmonary disease and emphysema),
  3. Diabetes (type I or II) that is not controlled with medication or diet,
  4. Hyperthyroidism,
  5. Uncontrolled seizures;
* Used any injection therapy (e.g., tender or trigger point injections, steroid injections), acupuncture, biofeedback, or TENS for the management of facial/jaw pain within 2 weeks prior to the screening assessment; If undergoing botulinum toxin injections in the head and neck area, must be 3 months since last set of injections and refrain from this treatment until study participation has ended
* History of major depression or other major psychiatric disorder requiring hospitalization within the last 6 months prior to the screening assessment;
* History of treatment for drug or alcohol abuse within the last 12 months;
* Current pain medication use (e.g., opioids, ibuprofen, acetaminophen) that cannot be stopped <24 hours prior to each study visit;
* Current use of medically prescribed muscle relaxants for the duration of study participation;
* Other conditions/diseases associated with altered pain perception: neurological or development disorders (dementia, autism spectrum disorder), neoplasm, multiple sclerosis, trigeminal neuralgia;
* Adults lacking capacity to provide informed consent for themselves;
* Unable to understand instructions for study procedures in English.
* Anything that would place the individual at increased risk or preclude the individual's full compliance with study procedures or completion of the study."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-01-12 (Estimated); Study Completion 2027-01-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of bad jaw pain fluctuations | 7 days following intervention
  Primary outcome includes the proportion of bad jaw pain fluctuations. A bad jaw pain fluctuation is defined as an increase ≥ 20 points from a previous measure. Jaw pain ratings will be collected daily for 8 days. The proportion of pain fluctuations is defined as the number of bad jaw pain fluctuations relative to the total number of jaw pain ratings.
Patient change in proportion of bad jaw pain fluctuations | 7 days following intervention
  Patient change in proportion of bad pain fluctuations will be assessed by comparing the proportion of bad jaw pain fluctuations between patients receiving heat therapy and matched patients not receiving heat therapy during the wait period.

CONTACTS AND LOCATIONS:
Overall Officials: Estephan Moana-Filho, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No